CLINICAL TRIAL: NCT01193062
Title: A Phase 1 Investigator And Subject-Blind Study In Healthy Subjects To Evaluate The Pharmacodynamic Effects Of Single Doses Of PF-04995274 On Sapp-Alpha Concentrations In Cerebrospinal Fluid Using Serial Sampling Methodology
Brief Title: Study In Healthy Subjects To Evaluate The Changes In The Protein sAPP-Alpha In Cerebrospinal Fluid Following A Single Oral Dose Of PF-04995274
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B1661004
Record Dates: First submitted 2010-08-25; First posted 2010-09-01 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: healthy volunteers; pharmacokinetics-pharmacodynamics; cerebrospinal fluid; serial sampling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects will be randomized to receive single oral doses of 0.1 mg, 10 mg, 15mg/ 40 mg PF-04995274 or a placebo
  Interventions: Drug: PF-04995274
- Cohort 2 (Experimental): Subjects will be receive single oral doses of PF-04995274 not exceeding 15mg or a placebo
  Interventions: Drug: PF-04995274

INTERVENTIONS:
Drug: PF-04995274 — Subjects will be randomized to receive single oral doses of 0.1 mg, 10 mg, 15mg/ 40 mg PF-04995274 or a placebo
  Arms: Cohort 1
Drug: PF-04995274 — Doses for cohort 2 will be decided based on an Interim analysis of data from cohort 1. The highest dose to be used in Cohort 2 not to exceed 15mg
  Arms: Cohort 2

SUMMARY:
The primary purpose of the study is to evaluate the effect of PF-04995274 on cerebrospinal fluid levels of soluble Amyloid precursor protein fragments and Amyloid beta fragments following single oral dose in healthy volunteers. Safety and tolerability of PF-04995274 single dose administration in healthy volunteers will also be assessed as part of the objectives.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the effect of PF-04995274 on CSF levels of s-APP and Abeta fragments following single oral dose in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* For all cohorts, healthy male and/or female subjects of nonchildbearing potential between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and heart rate measurement, 12 lead ECG and clinical laboratory tests).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing women; women of childbearing potential.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety Endpoints (AE's, Vital signs, ECG, Clinical safety laboratory endpoints, Clinical examinations) | duration of study
Cmax, Tmax, AUClast, AUCinf, and t1/2 of PF 04995274 and PF-05082547 in plasma, as the data permit | upto 5 days post dose
Cmax, Tmax, AUClast, AUCinf, and t1/2 of PF 04995274 and PF-05082547 in cerebrospinal fluid, as the data permit | upto 8 hrs post dose
Cmax, Tmax, AUClast, AUCinf, and t1/2 of s-APP alpha and Abeta fragments in cerebrospinal fluid, as the data permit | 8 hours post dose

SECONDARY OUTCOMES:
PK/PD model | 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1661004&StudyName=A%20Phase%201%20Investigator%20And%20Subject-Blind%20Study%20In%20Healthy%20Subjects%20To%20Evaluate%20The%20Pharmacodynamic%20Effects%20Of%20Single%20Doses%20Of%20PF-04995274%20On%20Sapp-Alpha%20Concentrations%20In%20Cerebrospinal%20Fluid%20Using%20Serial%20Sampling%20Methodology